CLINICAL TRIAL: NCT01014806
Title: A Phase 2a Randomized, Double-Blind, Active-Controlled Trial to Evaluate the Safety and Immunogenicity of a Trivalent Seasonal Influenza Virus-Like Particle (VLP) Vaccine (Recombinant) in Older Adults
Brief Title: Evaluate the Safety and Immunogenicity of a Seasonal Influenza Virus-Like Particle (VLP) Vaccine in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NVX755.202
Record Dates: First submitted 2009-11-14; First posted 2009-11-17 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose (Experimental)
  Interventions: Biological: Influenza VLP Vaccine
- High dose (Experimental): Investigational Influenza VLP Vaccine 60ug/strain
  Interventions: Biological: Influenza VLP Vaccine
- TIV (Active Comparator): Trivalent Influenza Vaccine 15ug/strain, Commercially Licenced
  Interventions: Biological: TIV

INTERVENTIONS:
Biological: Influenza VLP Vaccine — Single dose; 0.5mL
  Arms: High dose; Low dose
Biological: TIV — Trivalent Influenza Vaccine 15ug/strain, commercially licensed
  Arms: TIV

SUMMARY:
* To assess the tolerability and safety of a single injection of Influenza VLP Vaccine when administered intramuscularly (IM) at 15 µg and 60 µg HA per each strain.
* To assess the immunogenicity of Influenza VLP Vaccine administered at 15 µg and 60 µg HA per strain as measured by hemagglutination inhibition (HAI) antibody titers to each of the component viral strains [A/Brisbane/59/2007 (H1N1); A/Brisbane/10/2007 (H3N2) and B/Brisbane/60/2008].

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female > 60 years of age at the time of the vaccination.
2. Informed consent must be obtained from the subject prior to beginning any study specific procedures indicating that they understand the purpose of this study and are willing to adhere to the procedures described in this protocol.
3. Available by telephone.
4. Free of obvious health problems or chronic illnesses (i.e., recent exacerbation or acute episode of chronic illness in the last 3 months) as established by medical history, review of systems, and clinical examination before entering the study. This includes any mental condition that would interfere with subject self-assessment. Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable. Stable disease is defined as no new onset of exacerbation of pre-existing chronic disease 3 months prior to study vaccine injection.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
2. Receipt of any other licensed influenza vaccines or investigational influenza vaccine within 6 months prior to enrollment in this study or expected receipt of any vaccination before the final immune response blood collection.
3. History of hypersensitivity to any component of inactivated influenza vaccines, including egg or egg products, gelatin, or arginine.
4. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine. The use of inhaled and nasal steroids will be permitted.
5. Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
6. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.
7. Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever > 100.5F.
8. Acute clinically significant pulmonary, including asthma, cardiovascular, hepatic or renal functional abnormality as determined by physical examination or laboratory screening tests.
9. Major congenital defects that may increase the risk for influenza complications.
10. History of any neurological disorders or seizures (with the exception of febrile seizures during childhood) related to an underlying immune disease or disorder, such as but not limited to: multiple sclerosis, lupus, Guillain-Barre syndrome. Other neurological disorders that are clinically mild and stable with medication, such as mild Parkinson's disease, will not be excluded.
11. Any condition that in the opinion of the investigator would interfere with evaluation of the vaccine or interpretation of study results.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 0-21 days
Immunogenicity by HAI | 21 Days

SECONDARY OUTCOMES:
Immunogenicity by HAI compared to commercially licensed TIV vaccine | 21 days
Immunogenicity Against drifted strains by HAI | 21 days
Immunogenicity by neuraminidase activity inhibition (NAI) | 21 Days

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Universtity Clinical Research, Pembroke Pines, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Brown University, Providence, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Research Across America, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas